CLINICAL TRIAL: NCT07234539
Title: A Randomized Controlled Trial to Evaluate an Artificial Intelligence-enabled Clinical Assistant for Thyroid Cancer Staging and Risk Stratification Among Medical Students and Clinicians
Brief Title: Evaluation of an Artificial Intelligence-enabled Clinical Assistant to Support Thyroid Cancer Management
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Innovation and Technology Commission, Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Carlos King-Ho Wong, Honorary Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: UW24-319-RCT
Record Dates: First submitted 2025-09-29; First posted 2025-11-18 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-11

CONDITIONS: Thyroid Cancer; Large Language Models
Keywords: Thyroid Cancer; large language models; LLMs; natural language processing; NLP
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI-enabled clinical assistant (Experimental): Participants will provide the caner staging and risk category of each thyroid cancer patient as well as the participants' confidence for the above diagnostic assessments with AI-enabled clinical assistant as the intervention. The AI assistant is powered by LLMs and comprises a clinical dashboard. The clinical dashboard displays the original clinical notes and summarizes cancer staging and risk category of each thyroid cancer patient generated from the backend processing of the clinical assistant. Supporting evidence from original clinical notes is also highlighted for participants' verification.
  Interventions: Other: AI-enabled clinical assistant
- Manural chart review (No Intervention): Participants will provide the caner staging and risk category of each thyroid cancer patient as well as the participants' confidence for the above diagnostic assessments with manual chart review.

INTERVENTIONS:
Other: AI-enabled clinical assistant — Participants will provide the caner staging and risk category of each thyroid cancer patient as well as the participants' confidence for the above diagnostic assessments with AI-enabled clinical assistant as the intervention. The AI assistant is powered by LLMs and comprises a clinical dashboard. The clinical dashboard displays the original clinical notes and summarizes cancer staging and risk category of each thyroid cancer patient generated from the backend processing of the clinical assistant. Supporting evidence from original clinical notes is also highlighted for participants' verification.
  Arms: AI-enabled clinical assistant

SUMMARY:
This study aims to evaluate the clinical feasibility of adopting artificial intelligence (AI)-based models to improve clinical management of thyroid cancer.

DETAILED DESCRIPTION:
With recent advancements in technology, AI has become widely applicable to visual text recognition in clinical settings. AI-powered text recognition is emerging as a highly efficient, sustainable, and cost-effective tool for decision making and personalised medicine. Numerous studies have employed natural language processing (NLP) algorithms, particularly large language models (LLMs), to convert unstructured free-text from clinical consultation notes within electronic health records (EHR) into structured data, thus enriching individual clinical profiles in the EHR databases. Over time, these AI models have continuously improved their predictive accuracy and performance through self-learning (or unsupervised learning). While AI models had made a significant impact in oncology practices overseas, their utility for text recognition in oncology remains limited in Hong Kong. This proposed study aims to evaluate the clinical feasibility of adopting AI-based models to improve the end-user confidence in diagnostic accuracy and risk prediction using AI-assisted workflows in thyroid cancer management.

ELIGIBILITY:
Inclusion Criteria:

* medical students
* clinicians (including but not limited to surgeons, oncologists, pathologists)

Exclusion Criteria:

* medical students and clinicians who had reviewed the clinical notes or were involved in the processing of the clinical notes prior to the commencement of clinical experimental studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-10-02 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Cancer Staging and Risk Stratification by Participants Compared with Ground Truth across Intervention and Non-intervention Groups | Between intervention group and non-intervention group. Cross-over in 3-4 weeks
  The study will compare the accuracy of cancer staging and risk category assessed by the participants across the intervention group with AI assitance and non-intervention group without AI asssitance.
  The participants will review the clinical notes and assess the cancer staging and risk category for each thyroid cancer patient with or without the AI assistant. Participant provided assessments will be compared against the ground truth established by the clinical investigators of the study to guage the accuracy which is quantified as the percentage of correctly graded cancer staging and risk stratification. The accuracy will be compared between the intervention group and non-intervention groups using t-tests to evaluate the clinical impact of the AI assistant.
Participants' Confidence in Cancer Staging and Risk Stratification as Assessed by a 0-10 Scale Questionnaire | Between intervention group and non-intervention group. Cross-over in 3-4 weeks
  The study will compare the participants' confidence in grading cancer staging and risk category between the intervention group with AI assistance and non-intervention group without AI-assistance.
  After evaluating each thyroid cancer case for providing cancer staging and risk category, participants will complete a short questionnaire rating their confidence in providing their assessments on a scale from 0 (lowest) to 10 (hightest). Meanw confidence score will be compared between the intervention group and non-intervention group to evaluate the clinical impact of the AI assitant.
Efficiency | Between intervention group and non-intervention group. Cross-over in 3-4 weeks
  The time required to complete reviewing one set of clinical notes is compared between intervention and non-intervention groups

CONTACTS AND LOCATIONS:
Overall Officials: King Ho Carlos Wong, Principal Investigator — School of Public Health The University of Hong Kong; Man Him Matrix Fung, Principal Investigator — Department of Surgery, School of Clinical Medicine, The University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Department of Surgery, School of Clinical Medicine, The University of Hong Kong, Hong Kong
  - School of Public Health, The University of Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Only anonymized IPD used in results publications will be shared so that re-identification of individuals is not possible.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The IPD and supporting information will be available upon the completion of study (anticipated date as 31 December 2025) with results dissemination or publication, and will remain unending until required of removal.
Access Criteria: The IPD and supporting information will be available with results dissemination and publication as documents uploads or attachment. Anyone who has access to the articles will be able to access all the documents.

REFERENCES:
- [Result] Murphy GS, Szokol JW, Marymont JH, Avram MJ, Vender JS, Rosengart TK. Impact of shorter-acting neuromuscular blocking agents on fast-track recovery of the cardiac surgical patient. Anesthesiology. 2002 Mar;96(3):600-6. doi: 10.1097/00000542-200203000-00015. PMID 11873034